CLINICAL TRIAL: NCT00531726
Title: Investigation of Efficacy and Safety of Deep Brain Stimulation in Patients With Treatment Resistant Major Depression in a Multicenter, Double-blind, Prospectivly-designed Delayed-onset Study (Tiefe Hirnstimulation Zur Behandlung Therapieresistenter Depressionen-eine Multizentrische, Doppelblinde, Prospektive Studie Mit Einem Delayed-onset Design)
Brief Title: Berlin Deep Brain Stimulation Depression Study
Acronym: BDDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University Hospital Carl Gustav Carus (Other); Ludwig-Maximilians - University of Munich (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Malek Bajbouj, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDDS
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Sham Comparator)
  Interventions: Device: DBS of Cg25
- A (Experimental)
  Interventions: Device: DBS of Cg25

INTERVENTIONS:
Device: DBS of Cg25

SUMMARY:
In this study efficacy and safety of deep brain stimulation of the cingulate cortex in 20 patients with treatment resistant major depression will be investigated. In addition, the stress axis, the cortical GABAergic system, neurotrophins and event-related potentials will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patient is diagnosed with a severe major depressive episode
* patient is in a chronic current MDE and/or has had a history of recurrent MDEs
* patient has not had an acceptable clinical response due to failure with at least three antidepressant treatments during the current episode.
* patient has a score > 20 on the HAMD24
* patient is stable on current psychotropic medication for at least 6 weeks
* patient is >25 and <80 years
* Global Assessment of Function (GAF) score of < 45

Exclusion Criteria:

* Atypical Depression (according to DSM IV)
* Other relevant psychiatric axis I or axis II diseases
* Relevant neurological diseases
* Relevant cardiac or pulmonary diseases with enhances anaesthesiological risk (ASA Score > 3)
* Patient is currently enrolled in another investigational study not associated with the current study
* Patient has a history of, or evidence of, significant brain malformation or significant head injury
* Patient is likely to require a whole body MRI after implantation

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
HAMD/MARS score reduction | 4 weeks

SECONDARY OUTCOMES:
neurotrophic factor concentration, p300, cortical excitability measures, stress axis measures | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, Study Director — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitaetsmedizin Berlin, Berlin, Germany

REFERENCES:
- See also: contact: stimulation@charite.de — http://www.charite-psychiatrie.de/en/main/module/affektive-stoerungen.html